CLINICAL TRIAL: NCT02455778
Title: Effect of Intervention With Oral Cinnamon on Metabolic Profile and Body Composition of Asian Indians With Metabolic Syndrome in North India: A 16 Week Double Blind Placebo Control Trial
Brief Title: Effect of Oral Cinnamon Intervention in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Institute of Home Economics, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Cinnamon 2010
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinnamon (Experimental): 3 grams of oral cinnamon per day in form of capsules (6) along with standard diet and exercise protocol
  Interventions: Dietary Supplement: Cinnamon
- Placebo (Placebo Comparator): 2.5 grams of wheat flour per day in form of capsules ( 6) along with standard diet and exercise protocol
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cinnamon
  Arms: Cinnamon
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This double blind placebo control study with supplementation of oral Cinnamon is being conducted to test the hypothesis that in subjects with Metabolic Syndrome oral cinnamon may lead to improvement in body composition and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 25 -65 years
2. Subjects identified with any three of following:

   1. Fasting blood glucose ≥100 mg/ dL
   2. Waist circumference ≥ 90 cm ( males) ≥ 80 cm (females)
   3. Triglycerides ≥ 150 mg/dL
   4. High density lipoprotein cholesterol ≤ 40 mg/dL ( in males) , ≤ 50 mg/dL (in females)
   5. Blood pressure Systolic BP ≥ 130 mm Hg
   6. Diastolic BP ≥ 85 mm Hg
3. Subjects who were willing to participate in the study.
4. Subjects, if on medication for high blood pressure were stable and there was no change in the dosage for the past 3 months.

Exclusion Criteria:

1. Subjects suffering from other chronic diseases and metabolic complications such as cardiovascular disease, diabetes, renal disease, myocardial infarction and other endocrine disorders.
2. Subjects who were allergic to wheat flour and cinnamon.
3. Subjects who were on medication of anti dyslipidemic or hypoglycemic drugs.
4. Subjects who had undergone bypass procedure.
5. Subjects suffering from any debilitating disease such as tuberculosis, HIV etc.
6. Subjects suffering from uncontrolled hypothyroidism/ hyperthyroidism
7. Pregnant and lactating mothers

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | baseline to 4 months

SECONDARY OUTCOMES:
HbA1c | baseline to 4 months
Lipid profile | baseline to 4 months
Body fat percentage | baseline to 4 months
Blood pressure | baseline to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis-C-DOC Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, Delhi, India

REFERENCES:
- [Derived] Gupta Jain S, Puri S, Misra A, Gulati S, Mani K. Effect of oral cinnamon intervention on metabolic profile and body composition of Asian Indians with metabolic syndrome: a randomized double -blind control trial. Lipids Health Dis. 2017 Jun 12;16(1):113. doi: 10.1186/s12944-017-0504-8. PMID 28606084